CLINICAL TRIAL: NCT02150499
Title: A Safety and Tolerability Study of Levalbuterol Tartrate HFA Inhalation Aerosol Metered Dose Inhaler (MDI) in Pediatric Subjects Birth to ≤ 48 Months of Age With Reactive Airways Disease in an Acute Setting
Brief Title: A Study of Levalbuterol Tartrate HFA Inhalation Aerosol Metered Dose Inhaler (MDI) in Pediatric Subjects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP051-361
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-03

CONDITIONS: Asthma
Keywords: Acute Asthma exacerbation
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- levalbuterol tartrate HFA inhalation aerosol plus placebo HFA (Experimental): Three doses. Each dose comprised of 8 puffs (4 puffs of levalbuterol tartrate HFA inhalation aerosol 45 mcg/puff plus 4 puffs of placebo HFA) for 24 total puffs, cumulative dose of 540 mcg levalbuterol tartrate HFA inhalation aerosol
  Interventions: Drug: levalbuterol tartrate HFA inhalation aerosol; Drug: placebo
- levalbuterol tartrate HFA inhalation aerosol plus levalbuterol (Experimental): Three doses. Each dose comprised of 8 puffs (4 puffs of levalbuterol tartrate HFA inhalation aerosol 45 mcg/puff plus 4 puffs of levalbuterol tartrate HFA inhalation aerosol 45 mcg/puff) for 24 total puffs, cumulative dose of 1080 mcg levalbuterol tartrate HFA inhalation aerosol.
  Interventions: Drug: levalbuterol tartrate HFA inhalation aerosol

INTERVENTIONS:
Drug: levalbuterol tartrate HFA inhalation aerosol
  Other Names: Xopenex HFA® (Levalbuterol tartrate) Inhalation Aerosol
Drug: placebo
  Arms: levalbuterol tartrate HFA inhalation aerosol plus placebo HFA

SUMMARY:
This is a study of levalbuterol tartrate HFA inhalation aerosol MDI in pediatric subjects birth to ≤ 48 months of age who go to the Emergency Department (ED) or their physician's office with an acute bronchospasm. Subjects presenting to the ED or physician's office with an acute bronchospasm must have a history of reactive airways disease, based on subjects' parent/guardian report.

DETAILED DESCRIPTION:
This is a study to determine the safety and tolerability of cumulative dosing with levalbuterol tartrate HFA inhalation aerosol MDI using a valved holding chamber and facemask in pediatric subjects birth to ≤ 48 months of age with acute bronchospasm. It is a randomized, double-blind, parallel-group, multicenter, trial of 3 doses of levalbuterol tartrate HFA inhalation aerosol MDI in pediatric subjects birth to ≤ 48 months of age who present to either the Emergency Department (ED) or their physician's office with an acute bronchospasm. Subjects presenting to the ED or physician's office with an acute bronchospasm must have a history of reactive airways disease, based on subjects' parent/guardian report.

Eligible subjects whose parent(s) or legal guardian(s) provide written informed consent to participate will be randomized to 1 of 2 treatments. Treatment 1 consists of 3 doses, with each dose comprised of 8 puffs (4 puffs of levalbuterol tartrate HFA inhalation aerosol 45 mcg/puff plus 4 puffs of placebo HFA [cumulative dose of 540 mcg levalbuterol tartrate HFA inhalation aerosol]); Treatment 2 consists of 3 doses, with each dose comprised of 8 puffs of levalbuterol tartrate HFA inhalation aerosol 45 mcg/puff (4 puffs of levalbuterol tartrate HFA inhalation aerosol 45 mcg/puff plus 4 puffs of levalbuterol tartrate HFA inhalation aerosol 45 mcg/puff [cumulative dose of 1080 mcg of levalbuterol tartrate HFA inhalation aerosol]). For each Treatment, study medication will be administered every 20 minutes over a period of 1 hour for three doses.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female from birth to 48 months of age, inclusive, whose parent(s) or legal guardian(s) provide written informed consent prior to study participation and are willing to comply with study procedures.
2. Subject experiencing acute bronchospasm requiring a bronchodilator and who have a history of wheezing.

Exclusion Criteria:

1. Subject with a severe illness that, in the opinion of the Investigator, could jeopardize subject safety.
2. Subject received ≥ 8 puffs (MDI) of a beta-2 agonist or 2.5 mg of nebulized levalbuterol, or albuterol 5.0 mg within 4 hours prior to ED or physician's office admittance.
3. Subject received ipratropium within 4 hours prior to ED or physician's office admittance.
4. Subject who participated in an investigational drug study within 30 days prior to enrollment, or who previously participated in the current study.
5. Subject with a known sensitivity to levalbuterol or racemic albuterol or any of the excipients contained in any of these formulations.
6. Subject using any prescription drug (including beta-blockers) with which levalbuterol or racemic albuterol sulfate administration is contraindicated.
7. Subject with a history of clinically significant abnormalities that could interfere with the metabolism or excretion of the study medication (eg, renal, hepatic, metabolic, or endocrine abnormalities).
8. Subject with a history of cancer.

Max Age: 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Respiratory Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (17):
- United States (17):
  - Score Physician Alliance, LLC, St. Petersburg, Florida
  - Northern Illinios Research Associates, DeKalb, Illinois
  - Northern Illinois Associates, DeKalb, Illinois
  - Michael W. Simon, MD, PSC, Nicholasville, Kentucky
  - Willis-Knighton Physician Network / Portico Pediatrics, Shreveport, Louisiana
  - Mid Michigan Sleep Center, Grand Blanc, Michigan
  - Craig Spiegel, MD, Bridgeton, Missouri
  - St. Peter's University Hospital, New Brunswick, New Jersey
  - Capital Pediatrics & Adolescent Center PLLC, Raleigh, North Carolina
  - Capitol Pediatric & Adolescent Center PLLC, Raleigh, North Carolina
  - Dayton Clinical Research, Dayton, Ohio
  - Charleston Allergy & Asthma Research, Summerville, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - TTS Research, Boerne, Texas
  - Allergy Asthma Research Institute, Waco, Texas
  - PI-Coor Clinical Research, Burke, Virginia
  - Advanced Pediatrics, Vienna, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Levalbuterol Tartrate HFA Inhalation Aerosol Plus Placebo HFA: Three doses. Each dose comprised of 8 puffs (4 puffs of levalbuterol tartrate HFA inhalation aerosol 45 mcg/puff plus 4 puffs of placebo HFA) for 24 total puffs, cumulative dose of 540 mcg levalbuterol tartrate HFA inhalation aerosol
  levalbuterol tartrate HFA inhalation aerosol
  placebo
- Levalbuterol Tartrate HFA Inhalation Aerosol Plus Levalbuterol: Three doses. Each dose comprised of 8 puffs (4 puffs of levalbuterol tartrate HFA inhalation aerosol 45 mcg/puff plus 4 puffs of levalbuterol tartrate HFA inhalation aerosol 45 mcg/puff) for 24 total puffs, cumulative dose of 1080 mcg levalbuterol tartrate HFA inhalation aerosol.
  levalbuterol tartrate HFA inhalation aerosol
Period: Overall Study
Arm/Group | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Placebo HFA | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Levalbuterol
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pediatric subjects birth to less than or equal to 48 months of age with reactive airways disease in an acute setting
Groups:
- Total: Total of all reporting groups
Arm/Group | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Placebo HFA | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Levalbuterol | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 9 | 18
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 18.6 (10.21) | 17.1 (12.75) | 17.8 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: The Overall Safety of Treatment With Levalbuterol Tartrate HFA Inhalation Aerosol as Measured by the Number of Subjects With Treatment-emergent Adverse Events.
Description: Due to early termination of the study, insufficient data were available to perform the statistical analyses described in the protocol. Only subject listings of disposition, demographics, medical history and safety data were provided.
Time Frame: Week 1
Measure: Number; unit: Number of Adverse Events
Arm/Group | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Placebo HFA | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Levalbuterol
Number analyzed (Participants) | 9 | 9
Number of Adverse Events | 4 | 6

2. Primary Outcome: The Overall Safety of Treatment With Levalbuterol Tartrate HFA Inhalation Aerosol as Measured by the Number of Subjects With Serious Adverse Events.
Description: as for outcome 1
Time Frame: Week 1
Measure: Number; unit: Number of Serious Adverse Events
Arm/Group | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Placebo HFA | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Levalbuterol
Number analyzed (Participants) | 9 | 9
Number of Serious Adverse Events | 0 | 0

3. Primary Outcome: The Overall Safety of Treatment With Levalbuterol Tartrate HFA Inhalation Aerosol as Measured by the Number of Subjects With Treatment-emergent Adverse Events Leading to Discontinuation.
Description: as for outcome 1
Time Frame: Week 1
Measure: Number; unit: Number of Discontinuations
Arm/Group | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Placebo HFA | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Levalbuterol
Number analyzed (Participants) | 9 | 9
Number of Discontinuations | 0 | 0

4. Secondary Outcome: Change From Baseline in Pulmonary Score (Total Score) to End of Treatment
Description: as for outcome 1
Time Frame: Day 1
Arm/Group | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Placebo HFA | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Levalbuterol
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Pulmonary Score (Individual Component Scores) to End of Treatment
Description: as for outcome 1
Time Frame: Day 1
Arm/Group | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Placebo HFA | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Levalbuterol
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Pulmonary Score (Total Score) After Each Dose
Description: as for outcome 1
Time Frame: 20 minutes, 40 minutes, 60 minutes
Arm/Group | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Placebo HFA | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Levalbuterol
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Pulmonary Score (Individual Component Scores) After Each Dose
Description: as for outcome 1
Time Frame: 20 minutes, 40 minutes, 60 minutes
Arm/Group | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Placebo HFA | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Levalbuterol
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number and Percentage of Subjects Determined to be Stabilized After Treatment
Description: as for outcome 1
Time Frame: Day 1
Arm/Group | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Placebo HFA | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Levalbuterol
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: three months
Arm/Group | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Placebo HFA | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Levalbuterol
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 2/9 | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Placebo HFA (N=9) | Levalbuterol Tartrate HFA Inhalation Aerosol Plus Levalbuterol (N=9)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Existaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Termor (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish